CLINICAL TRIAL: NCT07018284
Title: Assessment of Postoperative Pain Incidence in Teeth Affected by Pulpitis, Necrosis, or Previously Treated, Following Obturation With Bioceramic or Resin-based Sealers
Brief Title: Postoperative Pain Evaluation After Obturation With Different Sealers
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Siena (Other)
Collaborators: Universidad Rey Juan Carlos (Other)
Responsible Party: Principal Investigator, Simone Grandini, Prof, University of Siena
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HSCO
Record Dates: First submitted 2025-06-04; First posted 2025-06-12 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-06

CONDITIONS: Periapical Periodontitis; Pulpitis; Necorsis
Keywords: Bioceramic sealers; Resin-based sealers; Endodontics
MeSH Terms: conditions — Periapical Periodontitis; Pulpitis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Active Comparator: AH Plus + Continuous Wave Condensation (Active Comparator): Root canal obturation using AH Plus (Dentsply Sirona, Charlotte, NC, USA) and the continuous wave technique with thermoplasticized gutta-percha
  Interventions: Procedure: AH Plus (Dentsply Sirona, Charlotte, NC, USA); Procedure: Continuous Wave Condensation
- Active Comparator: AH Plus + Single Cone (Experimental): Root canal obturation using AH Plus and the single cone technique with cold gutta-percha.
  Interventions: Procedure: AH Plus (Dentsply Sirona, Charlotte, NC, USA); Procedure: Single Cone Technique
- NeoSealer Flo + Continuous Wave (Experimental): Root canal obturation using NeoSealer Flo (Avalon Biomed, Houston, TX, USA) and the continuous wave technique.
  Interventions: Procedure: NeoSealer Flo; Procedure: Continuous Wave Condensation
- NeoSealer Flo + Single Cone (Experimental): Root canal obturation using NeoSealer Flo and the single cone technique.
  Interventions: Procedure: NeoSealer Flo; Procedure: Single Cone Technique

INTERVENTIONS:
Procedure: AH Plus (Dentsply Sirona, Charlotte, NC, USA) — Root canal obturation using AH Plus (Dentsply Sirona, Charlotte, NC, USA), a resin-based sealer with low solubility and shrinkage. Used in combination with gutta-percha for root canal filling
  Arms: Active Comparator: AH Plus + Continuous Wave Condensation; Active Comparator: AH Plus + Single Cone
Procedure: NeoSealer Flo — Root canal obturation using NeoSealer Flo (Avalon Biomed, Houston, TX, USA), a premixed bioceramic sealer based on calcium silicate. Used in combination with gutta-percha to enhance apical healing and biocompatibility.
  Arms: NeoSealer Flo + Continuous Wave; NeoSealer Flo + Single Cone
Procedure: Continuous Wave Condensation — A warm vertical compaction technique using heat-softened gutta-percha to obturate the canal in three dimensions. Considered the gold standard for achieving dense and homogenous root canal fillings.
  Arms: Active Comparator: AH Plus + Continuous Wave Condensation; NeoSealer Flo + Continuous Wave
Procedure: Single Cone Technique — A cold hydraulic condensation technique using a single gutta-percha cone matched to the last rotary file, combined with a high-flow sealer. Designed for simplified obturation with minimal operator variability
  Arms: Active Comparator: AH Plus + Single Cone; NeoSealer Flo + Single Cone

SUMMARY:
This study aims to evaluate the incidence and intensity of postoperative pain in patients undergoing root canal treatment on teeth diagnosed with pulpitis, pulp necrosis, or with previous endodontic treatment. Teeth will be obturated using either bioceramic or resin-based sealers. The primary objective is to determine whether the type of sealer significantly influences the level of postoperative pain as reported by patients. Pain intensity will be assessed using the Visual Analogue Scale (VAS) at three time points: immediately after treatment, 24 hours, and 72 hours postoperatively. The findings are expected to provide clinical insight into which obturation material may be more effective in minimizing postoperative discomfort.

ELIGIBILITY:
Inclusion Criteria:

Patients aged 18 years and older. Teeth with a diagnosis of pulpal necrosis or irreversible pulpitis. Informed consent provided for data usage.

Exclusion Criteria:

* Patients with systemic conditions that may impair healing (e.g., uncontrolled diabetes, immunosuppression).
* Asymptomatic presentation
* Teeth with root fractures, resorption, or open apices.
* Incomplete clinical or radiographic records.
* Cases with poor-quality radiographs or lack of standardization for evaluation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 270 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-01-30 (Estimated)

PRIMARY OUTCOMES:
Radiographic Success Based on Periapical Index (PAI) Criteria | Minimum 6 months after root canal treatment
  Radiographic outcome will be assessed using the Periapical Index (PAI) by Ørstavik et al. (1986), which categorizes periapical healing from 1 (normal periapical structures) to 5 (severe apical periodontitis). Success is defined as PAI scores of 1 or 2 (complete healing or healing in progress). Evaluations will be based on periapical radiographs (and CBCT when available) taken at follow-up after at least 6 months. The assessment will be performed by a calibrated blinded evaluator using reference radiographs.

SECONDARY OUTCOMES:
Clinical Success Based on Absence of Symptoms | Minimum 6 months after treatment
  Clinical success will be defined by the absence of pain, tenderness to percussion or palpation, swelling, mobility, and other signs of persistent infection. These parameters will be evaluated through standard clinical examination during follow-up visits.
Radiographic Success Based on CBCT Evaluation | Minimum 6 months after treatment
  When available, cone beam computed tomography (CBCT) images will be used to assess periapical healing. A modified periapical index (PAI-CBCT) will be used, evaluating the presence, size, and resolution of periapical radiolucencies. Lesion healing will be interpreted as success if there is full resolution or significant reduction in size compared to baseline.

CONTACTS AND LOCATIONS:
Overall Officials: José Aranguren, MsC, Study Director — Universidad Rey Juan Carlos , Madrid, Spain 28922; Simone Grandini, PhD, Principal Investigator — University of Siena
Locations (1):
- Universidad Rey Juan Carlos , Madrid, Spain 28922, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Undecided